CLINICAL TRIAL: NCT00361413
Title: An Investigator Initiated Double Blind Randomized Study of Alefacept Treatment Prevention of Graft Versus Host Disease in Myeloablative Stem Cell Transplantation
Brief Title: Alefacept for Prevention of Graft Versus Host Disease (GVHD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: company withdrawal of the drug
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Michael Shapira, MD, Hadassah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MYS-01-HMO-CTIL
Record Dates: First submitted 2006-07-31; First posted 2006-08-08 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2010-12

CONDITIONS: Graft Versus Host Disease
Keywords: Stem cell transplantation; GVHD; Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Alefacept; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Alefacept
  Interventions: Drug: Alefacept (AMEVIVE®)
- 2 (Placebo Comparator)
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Alefacept (AMEVIVE®) — Alefacept
  Other Names: Alefacept
  Arms: 1
Drug: control group — these patients will receive the same treatment as group A, without alefacept
  Arms: 2

SUMMARY:
Alefacept (AMEVIVE®) is an immunosuppressive dimeric fusion protein. It was shown to interfere with lymphocyte activation by specifically binding to the lymphocyte antigen, CD2, and inhibiting LFA-3/CD2 interaction. Alefacept was evaluated in two randomized, double-blind, placebo-controlled studies in adults with chronic (>1 year) plaque psoriasis and a minimum body surface area involvement of 10% who were candidates for or had previously received systemic therapy or phototherapy. The response to alefacept was significantly better in both studies. In both studies, onset of response to alefacept treatment (defined as at least 50% reduction of baseline Psoriasis Area and Severity Index (PASI)) began 60 days after the start of therapy.

Graft versus host disease (GVHD) is the most ominous side effect of allogeneic stem cell transplantation (SCT). It causes severe inflammatory process, which is usually located to the skin, gut and liver. Treatment of GVHD consists of various immuno-suppressive and immuno-modulating drugs, including steroids, cyclosporine, tacrolimus, methotrexate etc. These drugs unfortunately can also cause severe immunologic failure that makes the patient prone to infection and malignancy, and other medication-specific side effects. In spite of this effect on the immune system, not all of the patients achieve control of GVHD, which usually rapidly leads to death. Despite the use of innovative immunosuppressive modalities, the prognosis of steroid resistant GVHD is usually poor.

It was shown that CD2 depletion of allografts could prevent GVHD. Alefacept was never systemically tried in GVHD but A phase II study of BTI-322, a rat monoclonal IgG2b directed against the CD2 antigen in steroid-refractory acute GVHD showed a total response rate of 55%. We showed that alefacept might have a beneficial effect in controlling steroid resistant aGVHD and chronic GVHD. It was also shown to dramatically change the nature of transfusion associated GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 14-75 years old with a disease necessitating allogeneic SCT.
2. In order to increase security, only full matched donors will be allowed and must be willing and capable of donating peripheral blood stem cells preferably, or bone marrow progenitor cells using conventional techniques, and lymphocytes if indicated.
3. Patients must sign written informed consents.
4. Patients must have an ECOG PS ≤ 2; creatinine < 2.0 mg/dl; ejection fraction > 40%; DLCO > 50% of predicted; serum bilirubin < 3 gm/dl; elevated GPT or GOT > 3 x normal values.

Exclusion Criteria:

1. Not fulfilling any of the inclusion criteria.
2. Active life-threatening infection.
3. Overt untreated infection.
4. Hypersensitivity to alefacept.
5. HIV seropositivity, Hepatitis B or C antigen positivity with active hepatitis.
6. Pregnant or lactating women.
7. Donor contraindication (HIV seropositive confirmed by western blot).
8. Hepatitis B antigenemia.
9. Evidence of bone marrow disease.
10. Unable to donate bone marrow or peripheral blood due to concurrent medical condition.
11. Inability to comply with study requirements.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-06; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Acute GVHD occurrence. | 100d
Acute GVHD grading. | 100d

SECONDARY OUTCOMES:
Time to acute GVHD. | 100d
Chronic GVHD occurrence. | 180d
Chronic GVHD grading. | 180d
Engraftment/graft rejection. | 21d
Overall survival. | 180d
Disease free survival. | 180d
Infections. | 180d
Transplant-related mortality (TRM). | 180d
Immune reconstitution | 180d
Toxicity assessment according to the Common Terminology Criteria for Adverse Events (CTCAE) | 180d

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Department of Stem Cell Transplantation & Cancer Immunotherapy, Jerusalem, Israel

REFERENCES:
- [Background] Shapira MY, Resnick IB, Bitan M, Ackerstein A, Tsirigotis P, Gesundheit B, Zilberman I, Miron S, Leubovic A, Slavin S, Or R. Rapid response to alefacept given to patients with steroid resistant or steroid dependent acute graft-versus-host disease: a preliminary report. Bone Marrow Transplant. 2005 Dec;36(12):1097-101. doi: 10.1038/sj.bmt.1705185. PMID 16247429